CLINICAL TRIAL: NCT03396692
Title: PEF-Block & Ribs Fractures Effect of Posterior Exo-thoracic Fascia Block in the Pain Management of Ribs Fractures: a Prospective, Randomized Study
Brief Title: PEF-Block & Ribs Fractures
Acronym: PEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF 9860
Record Dates: First submitted 2017-12-15; First posted 2018-01-11 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Chest Trauma With Ribs Fractures
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (Active Comparator): Pain management use intravenous morphine patient-controlled analgesia (PCA)
  Interventions: Procedure: Intravenous morphine patient-controlled analgesia (PCA)
- Posterior exo-thoracic fascia block arm (Experimental): Pain management use intravenous morphine patient-controlled analgesia (PCA) and a block of the posterior exo-thoracic fascia with Ropivacaine
  Interventions: Procedure: Block of the posterior exo-thoracic fascia with Ropivacaine
- Paravertebral block arm (Experimental): Pain management use intravenous morphine patient-controlled analgesia (PCA) and a block of paravertebral space with Ropivacaine
  Interventions: Procedure: Block of paravertebral space with Ropivacaine

INTERVENTIONS:
Procedure: Intravenous morphine patient-controlled analgesia (PCA) — Group 1 control:
  * Morphine titration at 0.1 mg/kg
  * Establishment of PCA morphine:
  * concentration 1mg/ml
  * 1ml bolus
  * refractory period of 7 minutes
  * no maximum dose per day. Premedication of the patient with Ketamine 0.15 mg/kg and Propofol 0.5 mg /kg
  Arms: Control Arm
Procedure: Block of the posterior exo-thoracic fascia with Ropivacaine — Group 2 PEF block:
  * Establishment of PCA morphine:
  * concentration 1mg / ml
  * 1ml bolus
  * refractory period of 7 minutes
  * no maximum dose per day.
  * Realization of a block of the posterior exo-thoracic fascia (PEF block) at the median level of ribs fractures with ropivacaine 5mg / mL, 3 mg / kg under echography guidance. ALR needle (type neurostimulation) with a length of 100 mm is used. When the injection is performed an analgesia catheter is deposited in the space created by local anesthetics. Realization of ropivacaine bolus 2mg / ml at 0.1ml/kg every 4 hours. Possibility of an additional bolus of 0.1ml / kg every hour if insufficient analgesia.
  Arms: Posterior exo-thoracic fascia block arm
Procedure: Block of paravertebral space with Ropivacaine — Group 3 paravertebral block:
  * Establishment of PCA morphine:
  * concentration 1mg / ml
  * 1ml bolus
  * refractory period of 7 minutes
  * no maximum dose per day.
  * Realization of a paravertebral block (BPV) at the median level of ribs fractures ropivacaine 5mg / mL, (0.3ml / kg) 1.5 mg / kg under echography guidance. ALR needle (type neurostimulation) with a length of 100 mm is used. When the injection is performed an analgesia catheter is deposited in the space created by local anesthetics. Realization of bolus of ropivacaine 2mg / ml at 0.1ml / kg every 4 hours.
  Possibility of an additional bolus of 0.1ml / kg every hour if insufficient analgesia.
  In the case of failure of initial management with significant pain despite the iterative boli, epidural analgesia is used in recourse.
  Arms: Paravertebral block arm

SUMMARY:
Rib fractures are frequent injuries found approximately in 10% severe trauma patient. Rib fractures were correlated in many studies with a higher morbidity and mortality. This impaired outcome is mainly due to pulmonary complications consequences including especially pulmonary contusions. Frequently, patients present difficulty deep breathing and coughing. These adverse effects can lead to the development of atelectasis, hypoxia, and respiratory failure with mechanic ventilation recourse. Effective pain management may prevent these complications and reduce the likelihood of developing chronic pain. A multi-modal analgesia regimen is widely employed combining regional and systemic analgesia. Epidural analgesia is considered by many authors to be the gold standard of pain relief although many side-effects are frequently describe including hypotension, urinary retention nausea and vomiting. Paravertebral nerve blockade is an adequate alternative that provide similar quality of analgesia with lower incidence of complication. However, the failure rate associates with PVB is about 13% and it may be associated with hypotension (4.6%), accidental vascular puncture (3.8%), accidental pleural puncture (1.1%) and rarely pneumothorax (0.5%). Recently, a description of the intercostal paraspinal nerve block. This technic was performed for patients undergoing thoracic surgery without complications.More recently, a description of a new approach to provide thoracic analgesia named the Posterior Paramedian subchoroidal (PoPS) block. The authors consider this technique provide an analgesia of the anterior and the posterior branch of adjacent thoracic nerves. The investigators propose to investigate the effect of Posterior exothoracic fascial block.

ELIGIBILITY:
Inclusion Criteria:

* Major patients (18-80 years old)
* Affiliated to the social security
* Hospitalized following severe trauma associated with at least 2 unilateral ribs fractures
* EVA greater than or equal to 3 when coughing or when mobilizing care.
* Management of the patient in the first 24 hours post trauma.
* Patient not intubated.
* Collection of informed written consent, notification on the anesthesia sheet.

Exclusion Criteria:

* Minor patients,
* Patients under guardianship
* Pregnant or lactating women
* Allergy known to local anesthetics,
* Severe coagulopathy,
* Infection of the puncture site
* Neuromuscular pathology
* Chronic pain patients (long-term treatment with non-inflammatory steroidal, opioid, neuroleptic, antidepressant, antiepileptic),
* Intubated patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Consumption of opoïd | 24 hours

SECONDARY OUTCOMES:
cough pain intensity | 1 hour, 6hours, 12hours, 24hours

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Center, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramin S, Charbit J, Airoldi F, Courvallin E, Dagod G, Herteleer M, Choquet O, Bringuier S, Capdevila X. Continuous posterior extrathoracic fascial plane block versus continuous paravertebral block for pain management in patients with multiple rib fractures: a randomised controlled noninferiority trial. Br J Anaesth. 2025 Nov 20:S0007-0912(25)00735-4. doi: 10.1016/j.bja.2025.09.058. Online ahead of print. PMID 41271472